CLINICAL TRIAL: NCT01044615
Title: Advanced Imaging Tools in the Study of Mild Traumatic Brain Injury
Acronym: mTBI
Status: Completed | Type: Observational
Sponsor: Kettering Health Network (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: mTBI
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; Concussion; Magnetic Resonance Imaging (MRI); Positron Emission Tomography(PET); Computed Tomography (CT)
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild traumatic brain injury patients: Subjects who have a verifiable diagnosis of mild traumatic brain injury sustained within 24 months prior to enrollment
- Normal Control: Normal, healthy adults with no history of brain injury.

SUMMARY:
We will utilize a set of imaging modalities including computed tomography (CT), positron emission tomography (PET), and a suite of magnetic resonance imaging (MRI) tools, to investigate the changes in the human brain resulting from mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
We will recruit mTBI subjects and control subjects. Each subject will undergo the set of imaging modalities, and the results will be analyzed for differences at the structural, physiological, and molecular levels. The long term goal of this research is the development of a method to diagnose mTBI based on physical markers. This is a phased project beginning with a pilot study followed by future studies with larger sample sizes.

ELIGIBILITY:
Inclusion Criteria:

Study group:

* Between 18 and 55 years of age inclusive.
* Potential participant verbally verifies diagnosis of mTBI at pre-screen.
* Diagnosed with mild traumatic brain injury by a VAMC physician according to standard diagnostic criteria [12],[13], to be verified by chart review.
* Less than 24 months from trauma resulting in mTBI.
* Able to read and write in English.
* Willingness to refrain from nicotine, and beverages containing either alcohol or caffeine for at least four hours prior to the imaging session.
* Have signed the consent form for the study.

Control Group:

* Between 18 and 55 years of age inclusive.
* Potential participant verbally denies history of mTBI at pre-screen.
* Able to read and write in English.
* Willingness to refrain from nicotine, and beverages containing either alcohol or caffeine for at least four hours prior to the imaging session.
* Have signed the consent form for the study

Exclusion Criteria:

* Conditions that would preclude the completion of a MRI, PET, or CT exam such as claustrophobia, pacemaker, metal objects in body, and/or pregnancy.
* Serious, unstable medical or mental illness.
* Medical contraindication to any element of the study procedure.
* Have not read and signed an informed consent form, or do not understand its contents.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients at Veteran's Administration Medical Center in Dayton, OH who have history of Mild Traumatic Brain Injury within 24 months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Jason Parker, PhD, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Health Network, Kettering, Ohio, United States